CLINICAL TRIAL: NCT01667354
Title: Vaccine Hesitancy Intervention--Provider (VHIP)
Acronym: VHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Seattle Children's Hospital (Other); Washington State, Department of Health (Other Government); WithinReach (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 250147
Record Dates: First submitted 2012-03-06; First posted 2012-08-17 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Childhood Vaccination
Keywords: Parental Childhood Vaccine Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Clinics (Experimental): Providers in intervention clinics will receive a training followed by telephone coaching and follow-up visits for six months.
  Interventions: Behavioral: Academic Detailing
- Control Clinics (No Intervention): Control clinics will receive all intervention materials at the completion of the study.

INTERVENTIONS:
Behavioral: Academic Detailing — The intervention design is based on "academic detailing," an effective method of changing physician behavior. The aim of the training is effective communication with parents who are hesitant about childhood vaccinations.
  Arms: Intervention Clinics

SUMMARY:
The primary aim of this trial is to test the effectiveness of an intervention to train primary care physicians to determine if it leads to decreased parental vaccine hesitancy.

DETAILED DESCRIPTION:
The primary aim of this trial is to test the effectiveness of an intervention to train primary care physicians to determine if it leads to decreased parental vaccine hesitancy. The investigators will train primary care teams with an initial training followed by telephone coaching and follow-up visits, and assess the outcomes of parental vaccine hesitancy (primary) and physician self-efficacy (secondary) at baseline and 6 months.

ELIGIBILITY:
Study population:

* Eligible pediatric and family medicine practices in three counties in Washington State; King, Pierce and Snohomish Counties.
* Mothers whose infants will receive care in participating clinics.

Inclusion Clinics:

* Located in King, Snohomish, Pierce Counties, WA;
* Family practice clinics;
* Pediatric practice clinics;
* Order > 1000 doses of vaccine in 2009 from State of Washington Department of Health.

Exclusion Clinics: Not willing to be randomized.

Inclusion Mothers:

* Babies born at participating hospitals;
* Mother can be recruited before discharged post-birth;
* Mothers declare pediatric care at one of participating clinics;
* Singleton or twin pregnancies.

Exclusion Mothers:

* Babies born < 36 weeks gestational age;
* Known medical vaccine contraindications;
* Parental age < 18;
* NICU;
* Triplet or more;
* Maternal complications.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Parental Vaccine Hesitancy Measure | Change from Baseline in Parental Hesitancy at 6 months
  The investigators will contact mothers of newborns in study practices and conduct a telephone survey at two time points: baseline and 6 months. Surveys will assess parental hesitancy, parental trust in provider, and other covariates such as perceived social norms, other sources of information about vaccines, and demographic information.

SECONDARY OUTCOMES:
Physician Self Efficacy Measure | Change from Baseline in Physician Attitudes at 6 months
  Assessed via self-administered surveys of providers in all participating clinics at baseline and 6-months. The investigators will measure physician attitudes, perceived norms, intentions to change behavior, practice characteristics, and physician demographics.

CONTACTS AND LOCATIONS:
Overall Officials: David Grossman, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Henrikson NB, Opel DJ, Grothaus L, Nelson J, Scrol A, Dunn J, Faubion T, Roberts M, Marcuse EK, Grossman DC. Physician Communication Training and Parental Vaccine Hesitancy: A Randomized Trial. Pediatrics. 2015 Jul;136(1):70-9. doi: 10.1542/peds.2014-3199. Epub 2015 Jun 1. PMID 26034240